CLINICAL TRIAL: NCT04057560
Title: Metabolomics in Small Intestinal Bacterial Overgrowth
Acronym: MESIBO
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: United Lincolnshire Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 255049
Record Dates: First submitted 2019-07-23; First posted 2019-08-15 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Small Intestine Problem

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, urine, breath and mouth swabs, Small bowel fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SIBO Group
- Control Group

SUMMARY:
Small intestinal bacterial overgrowth (SIBO) is a condition where a person's own good and useful germs, live in parts of the bowel where there should not be any germs. It may cause difficult tummy and bowel symptoms in a wide variety of patient groups. Increasing evidence suggests that sometimes small intestinal bacterial overgrowth can also trigger or worsen diseases which do not have any bowel symptoms at all.

It is hugely under-diagnosed in clinical practice. Part of the reason for this is that current available diagnostic tests - culture of fluid sampled from the upper part of the gastrointestinal tract or breath testing, are complicated to do, difficult for the patient, and are not completely accurate. Therefore, the potential for a simple, more accurate test to revolutionise the diagnosis and aid with the treatment of this condition is immense.

When it is accurately diagnosed, treatment with antibiotics can cure the patient of their tummy or bowel symptoms.

Based on previous research the investigators have conducted, it is believed that it might be possible to diagnose this condition in a simpler and more accurate way by examining urine samples. This study will also investigate whether the condition could be diagnosed more accurately using a blood test, a different sort of breath test or using a mouth swab.

The proposed study will be conducted at Lincoln County Hospital, in collaboration with Joseph Banks Laboratory at the University of Lincoln. Additional urine, blood, swab and breath samples from patients with and without small intestinal bacterial overgrowth, before and after antibiotic treatment to identify specific molecular markers in urine, blood and saliva samples which diagnosis small intestinal bacterial overgrowth accurately.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged ≥ 18 and ≤ 50
2. Absence of red flag symptoms i.e. unexplained weight loss, a palpable mass, unexplained iron deficiency anaemia or rectal bleeding
3. GI symptoms which are due to possible SIBO
4. Capacity to give informed consent

Exclusion Criteria:

1. Presence of red flag symptoms (specified above in inclusion criteria)
2. Previous GI surgery including cholecystectomy (except appendicectomy, inguinal/femoral hernia repair or Caesarean sections)
3. Past history of inflammatory bowel disease, coeliac disease or pancreatic disease
4. Past history of cancer (except basal cell carcinoma)
5. Female patients who are pregnant
6. Inability to adequately understand verbal or written information
7. Inability or unwillingness to give informed consent
8. Unwilling to consider taking antibiotics to treat SIBO
9. Incapacity to comply with the demands of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients who are referred to Lincoln County Hospital for assessment of chronic diarrhoea will be considered eligible. They will be further assessed in a gastroenterology clinic using the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Metabolomic patterns in the biological samples collected from patients with SIBO | 12 months
  Metabolomic patterns in the biological samples collected from patients with SIBO
Metabolomic patterns in the biological samples collected from patients who do and do not report an improvement in clinical symptoms following antibiotic treatment | 12 moths
  Metabolomic patterns in the biological samples collected from patients who do and do not report an improvement in clinical symptoms following antibiotic treatment

SECONDARY OUTCOMES:
Changes in total Gastrointestinal Symptom Rating Scale scores in patients with SIBO before antibiotic treatment and following successful eradication of SIBO. | 12 months
  The Gastrointestinal Symptom Rating Scale is a self-assessed questionnaire consistsing of 32 individual gastrointestinal symptoms which are categorised into olfactory, upper GI, lower GI and anorectal subgroups. Each of the 32 items has a score of 0-3 (a high score represent a higher severity of the symptom). All 32 subscores will add up to give a total score.
Changes in stool types in patients with SIBO before antibiotic treatment and following successful eradication of SIBO. | 12 months
  This will be based on Bristol Stool Chart Type 1 to 7 stool (Type 1 is hard, lumpy stool and Type 7 is loose, watery stool)
Changes in improvement in quality of life in patients with SIBO before antibiotic treatment and following successful eradication of SIBO. | 12 months
  Quality of life of patients will be assessed using a visual analogue scale of 1 to 10 (higher values represent a better quality of life)

IPD SHARING:
Plan to Share IPD: No